CLINICAL TRIAL: NCT01514565
Title: Tumor Suppressor Status as a Predictor of Chemotherapy Response in Triple Negative Breast Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 11D-574
Record Dates: First submitted 2012-01-17; First posted 2012-01-23 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Triple negative Breast Cancer; RB; PTEN; Chemotherapy; Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective observational study aimed to validate biomarkers that predict response.

DETAILED DESCRIPTION:
This is a prospective observational cohort study, with no control group and no direct experimental intervention, where the patient's pathological material will be used to examine the expression of molecular biomarkers believed to predict chemotherapy response. Patients with locally advanced triple negative breast cancer, who are candidates for neoadjuvant chemotherapy, will be enrolled in this clinical study. Patients will receive standard of care, FDA-approved and clinically validated chemotherapy regimens. The biopsy specimens taken during the diagnostic phase (pre-treatment specimen) will be used for specific biomarker evaluation. Data obtained from this pre-treatment phase will be compared with the surgical specimens (post-treatment phase) obtained after receiving neoadjuvant chemotherapy. The primary endpoint is to assess the ability of specific biomarkers to predict treatment response, and thus identify those patients who will achieve benefit from such treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Histologically-confirmed triple negative invasive breast carcinoma
* Any type of ductal or lobular invasive carcinoma
* Patients with or without BRCA-1 and BRCA-2 mutations are eligible to participate
* Life expectancy > 6 months
* Pre-, Peri- or Postmenopausal
* Clinical Stage T2-4, N0-3, M0 (Stage II-III)
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial
* Adequate hematologic, renal, and liver function and functional status that permit chemotherapy administration. However, these parameters will be evaluated by the treating physician, and decisions regarding eligibility for chemotherapy or surgery will be made on a case by case scenario.

Exclusion Criteria:

* Prior history of and/or active therapy for invasive breast cancer (includes chemotherapy, radiation, hormonal therapy including AIs, tamoxifen, raloxifene, fulvestrant or any other antiestrogen/SERM)
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers are not to be registered. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are now considered to be at less than 30% risk for relapse (by their physician).
* Only ductal/lobular carcinoma in situ but not invasive component
* Any sort of confirmed metastatic disease (AJCC Stage IV at diagnosis)
* Any sort of active local radiation therapy (to the breast or the axilla), before the neoadjuvant chemotherapy
* Pregnant or lactating, in case this precludes the subject to receive chemotherapy.
* Impossibility to receive neoadjuvant chemotherapy due to significant medical comorbidities, allergies or performance status. This will be exclusively decided by the treating oncologists.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A maximum of 70 eligible patients will be enrolled. Accrual is expected to be completed in 18-24 months. All patients must have histologically confirmed triple negative breast cancer and be eligible to receive neoadjuvant chemotherapy.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Histological status of retinoblastoma tumour suppressor (RB) | Nine weeks
  The primary endpoint is to assess the impact of histological RB-status on pathological complete response (pCR). pCR is a well validated surrogate of chemotherapy sensitivity and allows the identification of a group of patients with excellent prognosis.

SECONDARY OUTCOMES:
Correlation of RB and other biomarkers | Nine weeks
  1. Correlation between RB and PTEN tumor suppressor status and other biomarkers with pCR
  2. Correlation between RB-status, RB and PTEN status and other biomarkers with recurrence free survival (RFS) and overall survival (OS)
Determine the utility of an RB molecular test | Assessed within 1 year
  Gene expression profiling of biopsy specimens to determine utility of an RB molecular test.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Witkiewicz, MD, Principal Investigator — Thomas Jefferson University; Gordon Schwartz, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States